CLINICAL TRIAL: NCT00892567
Title: Evaluation of CD8+ T Cell Activation and Infiltration Into Primary Breast Tumors Following Administration of a Peptide Vaccine
Brief Title: Evaluating the T Cell Response to a Peptide-based Vaccine in Patients With Breast Cancer
Acronym: Breast 37
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Craig L Slingluff, Jr (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Director, Human Immune Therapy Center, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12911; R21CA130340 (NIH)
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; peptide vaccine; immunotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 9 Peptide Vaccine (Experimental)
  Interventions: Biological: 9 Peptides from Her-2/neu, CEA, & CTA

INTERVENTIONS:
Biological: 9 Peptides from Her-2/neu, CEA, & CTA — Each vaccination will be administered on days 1, 8, 15, 36, 43, and 50. All participants will receive 9 class I MHC-restricted synthetic peptides and a class II MHC-restricted tetanus helper peptide administered in Montanide ISA-51. The vaccine will be administered subcutaneously (1 ml) and intradermally (1ml) at a single vaccination site.

SUMMARY:
The purpose of this study is to evaluate T cell responses against a peptide-based vaccine in patients with breast cancer and to determine whether peptide-specific T cells can be found at the site of breast tumors following vaccination.

DETAILED DESCRIPTION:
Just under 200,000 American women will be diagnosed with breast cancer this year. Standard breast cancer therapies have long included surgical resection, chemotherapy, radiation therapy, and hormonal therapy. However, other immune therapies are now being explored for the treatment of breast cancer, including peptide-based vaccines. In support of directed T cell therapies for breast cancer, antigenic epitopes from breast cancer-associated proteins such as Her-2/neu and the MAGE gene family have been identified, and vaccines containing peptides derived from these proteins have been shown to be safe and immunogenic in breast cancer patients.

Results from successful immune therapy approaches, for various human and murine cancers, have shown that antitumor effects can be mediated by T cells, which is proof-of-principle that the immune system, and in particular, T cells, can reject tumor. Overall, however, the complete clinical response rate for T cell mediated immunotherapies has been low. There are at least two possibilities to explain why this may be the case. First, tumor reactive T cells may not traffic to tumors. Second, tumor reactive T cells may not have adequate effector function within the tumor microenvironment. Neither of these hypotheses has been adequately explored, though there are data suggesting that either or both may represent obstacles to successful immune therapy. In order to improve upon the clinical response rate with vaccines, we need to address the questions of whether vaccine-induced T cells traffic to tumor and exhibit effector function within the tumor.

Specifically for breast cancer, there are opportunities for targeting T cells against primary tumors with the intent of providing immune protection early in the disease course. In the proposed clinical trial we will be administering a peptide-based vaccine and monitoring responses to the vaccine at the site of primary tumor. Peptide vaccines are unique in that they provide an opportunity to monitor directly the T cell response to defined antigens, enabling dissection of the immune response pre- and post-vaccination. The proposed analyses are designed to test the hypotheses that vaccination 1) enhances T cell infiltration into tumor and 2) induces T cells to become activated and fully differentiate into effector cells. The goals of this proposal are to define the extent to which these two processes occur following vaccination and to identify opportunities for improving tumor targeting and T cell effector function in human breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a mass approximately ≥1 cm by breast imaging, BIRADS 5
2. Patients who have been diagnosed, by cytologic or histologic examination, with adenocarcinoma (including invasive lobular carcinoma) of the breast and have not yet undergone primary surgery for their disease.
3. All participants must have:

   * ECOG performance status of 0 or 1
   * Ability and willingness to give informed consent
4. Laboratory parameters as follows:

   * HLA-A1, -A2, -A3, or -A31 (+)
   * ANC > 1000/mm3
   * Platelets > 100,000/mm3
   * Hgb > 11 g/dL
   * HGBA1C < 7%
   * AST and ALT ≤ 2.5 x upper limits of normal (ULN)
   * Bilirubin ≤ 2.5 x ULN
   * Alkaline phosphatase ≤ 2.5 x ULN
   * Creatinine ≤ 1.5 x ULN
   * HIV negative
   * Hepatitis negative
5. Age ≥ 18 years at the time of registration
6. Participants must have an intact (undissected), nodal basin in the upper extremity opposite the site of tumor.

Exclusion Criteria:

1. Patients who require neoadjuvant chemotherapy prior to surgery for the treatment of their disease.
2. Participants with known or suspected allergies to any component of the vaccine.
3. Participants who have an active infection requiring antibiotics.
4. Participants receiving the following medications or treatments at study registration or within the preceding 30 days are excluded:

   * Surgery
   * Chemotherapy
   * Radiation therapy
   * Allergy desensitization injections
   * Systemic corticosteroids, administered parenterally or orally. Inhaled steroids (e.g. Advair®, Flovent®, Azmacort®) are not permitted. Topical corticosteroids are acceptable, including steroids with very low solubility administered nasally for local effects only (e.g. Nasonex®).
   * Growth factors (e.g., Procrit®, Aranesp®, Neulasta®)
   * Any investigational medication
5. Participants may not have been vaccinated previously with any of the synthetic peptides included in this protocol.
6. Pregnancy during vaccine administration. Female participants of childbearing potential must have a negative pregnancy test (urinary or serum β-HCG) prior to administration of the first vaccine dose. Males and females must agree, in the consent form, to use effective birth control methods during the course of vaccination.
7. Female participants must not be breastfeeding.
8. Participants in whom there is a medical contraindication or potential problem in complying with the requirements of the protocol, in the opinion of the investigator.
9. Participants classified according to the New York Heart Association classification as having Class III or IV heart disease.
10. Participants must not have had prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement. Participants with an active autoimmune disorder requiring these therapies are also excluded. The following will not be exclusionary:

    * The presence of laboratory evidence of autoimmune disease (e.g. positive ANA titer) without symptoms
    * Clinical evidence of vitiligo
    * Other forms of depigmenting illness
    * Mild arthritis requiring NSAID medications
11. Body weight < 110 lbs (without clothes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To evaluate whether a multi-peptide vaccine induces T cells that traffic to and penetrate into human primary breast cancers. | 22 days following initiation of the vaccines

SECONDARY OUTCOMES:
To characterize the T cell response to a peptide-based vaccine in terms of antigen specificity and the induction of differentiated effector cells, both in the peripheral blood and within the tumor microenvironment. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David R. Brenin, M.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States